CLINICAL TRIAL: NCT05461924
Title: The Long Term Outcomes After Pull-through of Long Segment Hirschsprung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weibing Tang (Other)
Responsible Party: Sponsor-Investigator, Weibing Tang, Doctor, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Other Study IDs: NanjingCH-01
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Constipation; Incontinence; Hirschsprung Disease, Long-Segment; Long Term Adverse Effects
Keywords: Hirschsprung disease associated enterocolitis; bowel function
MeSH Terms: conditions — Constipation; Hirschsprung Disease; Long Term Adverse Effects | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- long-segment HSCR: Aganglionosis of non-rectosigmoid HSCR can extend to the descending colon, transverse colon, ascending colon, but not to the terminal ileum
  Interventions: Other: questionnaire survey
- rectosigmoid HSCR: Aganglionosis confined to the rectosigmoid
  Interventions: Other: questionnaire survey

INTERVENTIONS:
Other: questionnaire survey — questionnaire survey the long term outcomes of long-segment HSCR and compared with rectosigmoid HSCR

SUMMARY:
Hirschsprung disease (HSCR) is characterized by the absence of ganglion cells (aganglionosis) in the distal bowel extending proximally for varying distances that results in persistent spasm in the affected bowel and functional intestinal obstruction. Patients can be classified as rectosigmoid HSCR when aganglionosis confined to the rectosigmoid and long-segment or total colonic HSCR when aganglionosis extends beyond the upper sigmoid. Aganglionosis of long-segment HSCR can extend to the descending colon, transverse colon, ascending colon, but not to the terminal ileum. To date, there is insufficient evidence to recommend a preferred or superior method for the surgical repair for long-segment HSCR. In general, a pull-through with standard of care for the intestine and mesentery, which avoids excessive resection of the colon and coloanal reconstruction, is performed for long-segment HSCR.There are reports that a significant percentage of long-segment HSCR patients continue to have difficulty with soiling and incontinence,however there were also reports long-segment HSCR patients have the same continece as rectosigmoid HSCR.The outcome of long-segment HSCR should be thoroughly evaluated. The present study was designed to evaluate the long-term outcomes of long-segment HSCR.

DETAILED DESCRIPTION:
Hirschsprung disease (HSCR) is characterized by the absence of ganglion cells (aganglionosis) in the distal bowel extending proximally for varying distances that results in persistent spasm in the affected bowel and functional intestinal obstruction. Patients can be classified as rectosigmoid HSCR when aganglionosis confined to the rectosigmoid and long-segment or total colonic HSCR when aganglionosis extends beyond the upper sigmoid. Aganglionosis of long-segment HSCR can extend to the descending colon, transverse colon, ascending colon, but not to the terminal ileum. To date, there is insufficient evidence to recommend a preferred or superior method for the surgical repair for long-segment HSCR. In general, a pull-through with standard of care for the intestine and mesentery, which avoids excessive resection of the colon and coloanal reconstruction, is performed for long-segment HSCR.There are reports that a significant percentage of long-segment HSCR patients continue to have difficulty with soiling and incontinence,however there were also reports long-segment HSCR patients have the same continece as rectosigmoid HSCR.The outcome of long-segment HSCR should be thoroughly evaluated. The present study was designed to evaluate the long-term outcomes of long-segment HSCR.

The long-term outcome would be indicated by bowel function SCORE.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Hirschsprung disease Must be performed with the operation of pull-through Must be followed up more than 3 years

Exclusion Criteria:

Clinical diagnosis of Down syndrome Clinical diagnosis of tolal colonic Hirschsprung disease Clinical diagnosis of degestive malformation except Hirschsprung disease

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with with rectosigmoid and long-segment Hirschsprung disease after operation.
  The follow-up age must more than 3 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Bowel function score | through study completion, an average of 5 year
  Bowel function was evaluated by the BFS (20 points), which was approved by Rintala in 1995 ; patients with a score > 18 were considered to have normal bowel habits.

SECONDARY OUTCOMES:
Hirschspurng disease associated entrocolitis(HAEC) | through study completion, an average of 5 year
  The guidelines for the diagnosis and management of HAEC were defined by the American Pediatric Surgical Association in 2017

CONTACTS AND LOCATIONS:
Overall Officials: Changgui Lu, Dr, Principal Investigator — Department of pediatric surgery of Children's hospital of Nanjing medical unverisity
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No